CLINICAL TRIAL: NCT04819906
Title: A Randomized, Placebo- and Active-controlled 4-way Crossover Study in Healthy Subjects to Evaluate the Effect of E4 on the QTc Interval
Brief Title: Effect of Estetrol Monohydrate (E4) on QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIT-Do001-C104
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Prolonged QTc Interval
Keywords: Estetrol; Moxifloxacin
MeSH Terms: interventions — Estetrol; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- T-ST-P-M (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- ST-M-T-P (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- P-T-M-ST (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- M-P-ST-T (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- ST-P-T-M (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- P-M-ST-T (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- T-ST-M-P (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- M-T-P-ST (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- P-T-ST-M (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- T-M-P-ST (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- ST-P-M-T (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg
- M-ST-T-P (Experimental): Treatment T: Therapeutic E4 dose (20 mg): one E4 20 mg tablet plus four E4 placebo tablets
  Treatment ST: Supratherapeutic E4 dose (100 mg): five E4 20 mg tablets
  Treatment P: Placebo: five E4 placebo tablets
  Treatment M: Moxifloxacin: 1 moxifloxacin 400 mg tablet
  Interventions: Drug: Estetrol 20 mg; Drug: Estetrol 100 mg; Drug: Placebo; Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Estetrol 20 mg — One estetrol monohydrate (E4) 20 mg tablet plus four matching placebo tablets orally once
  Other Names: E4 20 mg
Drug: Estetrol 100 mg — Five estetrol monohydrate (E4) 20 mg tablets orally once
  Other Names: E4 100 mg
Drug: Placebo — Five placebo tablets orally once
Drug: Moxifloxacin 400 mg — One moxifloxacin 400 mg tablet orally once (open-label)

SUMMARY:
The purpose of this study is:

* to evaluate if E4 has any effect on how the heart beats when a single dose is given at two different dose levels;
* to determine the ability to detect small changes in how the heart beats using a positive control: moxifloxacin, a quinolone antibiotic approved by the FDA as a positive control in thorough QT (TQT) studies;
* to assess the safety and tolerability of a single dose of E4 administered at two different dose levels;
* to measure the amount of study drug in the blood stream and how long it takes for the body to eliminate it (Pharmacokinetics) after administration.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, randomized, placebo- and active-controlled, partially double-blinded, single-dose, 4-way crossover study in healthy postmenopausal female participants to evaluate the effect of E4 on the QTc interval. All participants will receive all 4 study treatments (E4 therapeutic dose [20 mg]; E4 supratherapeutic dose [100 mg]; placebo; moxifloxacin [400 mg]) in a randomized sequence.

E4 and placebo administration will be blinded while moxifloxacin will be provided in an open-label fashion.

Participants will report to the clinical research unit (CRU) for the eligibility screening within 28 days prior to the first study drug administration. Participants will sign the study specific informed consent form (ICF) prior to any study specific screening procedures being performed.

In each study period, the participants will be confined in the CRU from the day before dosing (Day -1) until all safety assessments have been completed on Day 2, for a total of 2 days per period. Each study period will be separated by a 14 day (±2 days) washout.

Cardiodynamic assessment using continuous 12-lead ECG (Holters) recordings will be performed on Day 1 of each treatment period starting approximately 1 hour before dosing and ending approximately 25 hours after dosing. ECGs will be extracted serially pre- and postdose and at predefined time points. Blood draws for PK will be performed in all periods after each ECG extraction.

All participants (including participants who terminate the study prematurely) will receive a follow-up call 7 (±2) days after the last administration of study treatment to determine if any adverse events (AEs) have occurred since the last study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, postmenopausal women, 40 years to 65 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose of study drug.
3. Minimum weight of 52 kg and body mass index (BMI) ≥18.0 and ≤32.0 kg/m2 at screening.
4. Healthy status defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including gynecological examination, vital signs, a 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology, and urinalysis clinical laboratory tests.
5. Postmenopausal status will be defined as any of the following:

   1. For non-hysterectomized participants:

      * at least 12 months of spontaneous amenorrhea; or
      * at least 6 months of spontaneous amenorrhea with serum FSH >40 mIU/mL (value obtained after washout of estrogen/progestin containing drugs, see exclusion criteria 18 and 20); or
      * at least 6 weeks postsurgical bilateral oophorectomy.
   2. For hysterectomized participants:

      * serum FSH >40 mIU/mL (values obtained after washout of estrogen/progestin containing drug, see exclusion criteria 18 and 20); or
      * at least 6 weeks postsurgical bilateral oophorectomy.
6. Understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the protocol.
7. Supine or semi-recumbent blood pressure between 90/40 mmHg and 150/90 mmHg (inclusive) at screening.
8. No clinically significant history or presence of 12-lead ECG findings as judged by the Principal Investigator at screening and check-in, including each criterion as listed below:

   * normal sinus rhythm (heart rate between 40 bpm and 100 bpm, inclusive).
   * Fridericia-corrected QTc (QTcF) interval ≤450 msec.
   * QRS interval ≤120 msec; and confirmed by manual over read if >120 msec.
   * PR interval ≤220 msec.
9. Has serum potassium, calcium, and magnesium levels within the normal range at screening.
10. Ability and willingness to abstain from alcohol-, caffeine-, and xanthine-containing beverages or food (eg, coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) before each admission to the clinical research unit (CRU) until clinic discharge.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Principal Investigator.
2. History of any illness that, in the opinion of the Principal Investigator, might confound the results of the study or pose an additional risk to the participant by their participation in the study.
3. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose of study drug.
4. History or presence of hypersensitivity or idiosyncratic reaction to E4, moxifloxacin, related compounds, or inactive ingredients.
5. History of significant multiple and/or severe allergies (e.g., latex allergy, band aids, adhesive dressing, or medical tape), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs.
6. Positive urine drug or alcohol results at screening or check-in.
7. Positive results at screening for human immunodeficiency virus (HIV), syphilis, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Unable to refrain from or anticipates the use of:

   * any drug, including prescription and nonprescription medications (including antacids), herbal remedies, or vitamin supplements (especially those containing magnesium, aluminum, iron, or zinc; exception: vitamin C may be allowed) beginning 14 days before the first dose of study drug and throughout the study; or
   * any drugs known to be significant inhibitors or inducers of cytochrome P450 (CYP) enzymes and/or P-glycoprotein (P-gp), including St. John's wort, for 28 days before the first dose of study drug and throughout the study. Appropriate sources will be consulted by the Principal Investigator or designee to confirm lack of pharmacokinetic (PK) or pharmacodynamic interaction with the study drug.
9. Has been on a diet incompatible with the on-study diet (including an extreme diet which resulted in a significant weight change for whatever reason), in the opinion of the Principal Investigator, within 28 days before the first dose of study drug, and throughout the study.
10. Donation of blood or significant blood loss more than 500 mL within 56 days before the first dose of study drug.
11. Plasma donation within 7 days before the first dose of study drug.
12. Has had surgery or any medical condition which may affect the absorption, distribution, metabolism, or elimination of the study drug within 6 months before the first dose, in the opinion of the Principal Investigator. Cholecystectomy is not exclusionary unless participant has post-cholecystectomy diarrhea.
13. Participation in another clinical study within 28 days before the first dose of study drug. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
14. Participation in a previous clinical study where participant received E4 <8 weeks after last dose of study drug.
15. Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
16. Strenuous activity, sunbathing, and contact sports within 48 hours (2 days) prior to admission to the CRU and for the duration of the study.
17. History or presence of:

    * clinically significant hypokalemia, in the opinion of the Principal Investigator; or
    * risk factors for Torsades de Pointes (eg, heart failure, cardiomyopathy, or family history of Long QT Syndrome); or
    * sick sinus syndrome, second, or third degree atrioventricular block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QTc interval, or conduction abnormalities; or
    * repeated or frequent syncope or vasovagal episodes; or
    * clinically significant cardiovascular disorders such as hypertension or bradycardia, or severe peripheral arterial circulatory disorders.
18. Use of estrogen/progestin containing drug(s) up to:

    * 1 week before screening for vaginal non-systemic hormonal products (rings, creams, gels); or
    * 4 weeks before screening for vaginal or transdermal estrogen or estrogen/progestin products; or
    * 8 weeks before screening for oral estrogen and/or progestin products and/or selective ER modulator therapy; or
    * 8 weeks before screening for intrauterine progestin therapy.
19. Use of androgen or dehydroepiandrosterone (DHEA)-containing drugs: 8 weeks before screening start for oral, topical, vaginal, or transdermal androgen.
20. Use of estrogen/progestin- and androgen/DHEA-containing drug(s) requiring a pre-screening washout longer than 8 weeks (progestin implants or estrogen alone injectable drug therapy, estrogen pellet therapy, or progestin injectable drug therapy, implantable, or injectable androgen therapy).
21. History of malignancy, with the exception of basal cell or squamous cell carcinoma of the skin if diagnosed more than 1 year before the screening visit.
22. Any clinically significant findings found by the Investigator at the breast examination and/or on mammography suspicious of breast malignancy that would require additional clinical testing to rule out breast cancer (however, simple cysts confirmed by ultrasound are allowed). Breast Imaging Reporting and Data System (BI-RADS) score other than 1 or 2 on mammogram.
23. Abnormal cervical Pap smear in non-hysterectomized participants with evidence of cervical dysplasia greater than low-grade squamous intraepithelial lesion (LSIL). Women with a diagnosis of atypical squamous cells of undetermined significance (ASCUS) may be enrolled. Pap smears will not be required for non-hysterectomized participants who have written documentation of prior test within 3 years.
24. For non-hysterectomized participants:

    * history or presence of uterine cancer, endometrial hyperplasia, disordered proliferative findings; or
    * presence of endometrial polyps; or
    * undiagnosed vaginal bleeding or undiagnosed abnormal uterine bleeding; or
    * endometrial ablation; or
    * any uterine/endometrial abnormality that, in the judgment of the Investigator, contraindicates the use of estrogen therapy. This includes presence or history of adenomyosis or significant myoma.
25. History or presence of venous or arterial thromboembolic disease (eg, deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, angina pectoris, etc.) or history of known coagulopathy.
26. Contraindications for the use of steroids for menopausal hormonal therapy at the investigator's discretion.
27. Participants who are not in euthyroid condition (hyperthyroidism or hypothyroidism), including participants who receive drug treatment (eg, L-thyroxine or anti-thyroid drugs).
28. Positive pregnancy test result at screening or Day -1.
29. Employee of PRA, the CRU, or the Sponsor.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Effect of E4 20 mg and E4 100 mg on QTc interval: placebo-corrected change from baseline QTcF (ΔΔQTcF) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).

SECONDARY OUTCOMES:
Effect of E4 20 mg and E4 100 mg on heart rate (HR): change-from-baseline heart rate (∆HR) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).
Effect of E4 20 mg and E4 100 mg on heart rate (HR): placebo-corrected change-from-baseline heart rate (∆∆HR) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).
Effect of E4 20 mg and E4 100 mg on PR interval: change-from-baseline PR interval (∆PR) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).
Effect of E4 20 mg and E4 100 mg on PR interval: placebo-corrected change-from-baseline PR interval (∆∆PR) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).
Effect of E4 20 mg and E4 100 mg on QRS duration: change-from-baseline QRS duration (∆QRS) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).
Effect of E4 20 mg and E4 100 mg on QRS duration: placebo-corrected change-from-baseline QRS duration (∆∆QRS) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECG time points (-45, -30, and -15 minutes).
Sensitivity Assay: effect of moxifloxacin 400 mg on QTc interval: placebo-corrected change from baseline QTcF (ΔΔQTcF) | from 45 minutes pre-dose to 24 hours post-dose
  Continuous 12-lead ECG (Holters) recordings will be performed. Baseline will be the average of the derived ECG intervals from the 3 predose ECGs extracted at -45, -30, and -15 minutes.
Frequency of Adverse events (AEs), Treatment-emergent adverse events (TEAEs), and Serious adverse events (SAEs) | from Day -1 of Period 1 up to end of study (i.e. 7 (±2) days after the last dose of study drug)
  Any clinically significant observations, as determined by the Investigator, in results of clinical laboratory tests, 12-lead ECGs, vital sign measurements, or physical examination findings will be recorded as Adverse events (AEs). At several time points before and after study drug administration, participants will be asked nonleading questions to determine the occurrence of AEs. In addition, all AEs reported spontaneously during the course of the study will be recorded.
  A treatment-emergent AE (TEAE) is defined as any event not present prior to the first administration of the study drug or any event already present that worsens in either severity or frequency following exposure to the study drug.
Maximum observed plasma concentration (Cmax) for E4 | from 1 hour pre-dose to 24 hours post-dose
Time to attain maximum observed plasma concentration (tmax) for E4 | from 1 hour pre-dose to 24 hours post-dose
Area under the plasma concentration-time curve up to 24 hours (AUC0-24) for E4 | from 1 hour pre-dose to 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Miami, Miami, Florida, United States